CLINICAL TRIAL: NCT00293501
Title: A Phase I/II Trial of Tinzaparin (Innohep), a Low Molecular Weight Heparin (LMWH) for Treatment of Advanced Renal Cell Carcinoma
Brief Title: Tinzaparin in Treating Patients With Metastatic Kidney Cancer That Cannot Be Removed By Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Vermont (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000459794; VCC-0403; VCC-05-040
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2007-02

CONDITIONS: Kidney Cancer
Keywords: clear cell renal cell carcinoma; stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Tinzaparin

INTERVENTIONS:
Drug: tinzaparin sodium

SUMMARY:
RATIONALE: Tinzaparin may stop the growth of kidney cancer by blocking blood flow to the tumor.

PURPOSE: This phase I/II trial is studying the side effects of tinzaparin and to see how well it works in treating patients with metastatic kidney cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effect of tinzaparin sodium on fibrin formation (prothrombin fragment F1.2), thrombin generation (thrombin-antithrombin complexes), and fibrinolysis (D-Dimer) from baseline to 2 weeks and at nadir or disease progression in patients with unresectable metastatic renal cell carcinoma (RCC).

Secondary

* Determine the effect of tinzaparin sodium treatment on circulating angiogenesis markers, including vascular endothelial growth factor (VEGF) and basic fibroblast growth factor (bFGF).
* Determine the proportion of patients developing venous thromboembolism and hemorrhage.
* Determine the tolerability of tinzaparin sodium treatment for up to 6 months in these patients.
* Establish the feasibility of undertaking a multicenter renal cell carcinoma trial with specialized coagulation test collection, shipping, and processing.
* Obtain more accurate and specific mean, median, and variability in biomarker data in advanced RCC patients treated with tinzaparin sodium for purposes of planning larger future trials.
* Estimate the progression-free survival at 4 months in patients treated with tinzaparin sodium.
* Correlate progression-free survival with changes in markers of coagulation activation or angiogenesis.
* Correlate the anticoagulant activity of tinzaparin sodium (anti-Xa activity) with change in coagulation markers, angiogenesis markers, and progression-free survival.

OUTLINE: This is an open-label, pilot, multicenter study.

Patients receive a treatment dose of tinzaparin sodium subcutaneously (SC) once daily for 14 days followed by a prophylactic dose of tinzaparin sodium SC once daily for up to 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed renal cell carcinoma of clear cell histology

  * Tumors of mixed histology eligible if ≥ 50% of tumor has clear cell histology
  * No nonclear cell histologies, collecting duct tumors, oncocytomas, or transitional cell tumors
* Metastatic and unresectable disease that is clinically extending beyond the regional lymph nodes (histological confirmation not required)

  * Patients who are inoperable for their primary tumor representing the sole site of disease are ineligible
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 2 cm by conventional techniques OR ≥ 1 cm by spiral CT scan
* No known brain metastases

PATIENT CHARACTERISTICS:

* Expected survival > 2 months
* CALGB (ECOG/ZUBROD) performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Hemoglobin ≥ 10 g/dL
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST/ALT ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN
* INR ≤ 1.5 times control value
* PTT < 1.5 times control value
* Negative pregnancy test
* Fertile patients must use effective contraception
* Patients must be able to receive subcutaneous injections at home
* No other primary malignancy in the past 5 years other than basal cell carcinoma or carcinoma in situ of the cervix that has been curatively treated and is associated with a less than 30% risk of relapse in the next 5 years
* No signs or symptoms of bleeding within 4 the past weeks
* No known bleeding diathesis or high risk for bleeding due to any condition, including trauma within the past 4 weeks, active current bleeding, or hemorrhagic stroke or intraocular bleeding within the past 6 months
* No active thromboembolism highly likely to require anticoagulation during the study period
* No known or suspected history of type II heparin-induced thrombocytopenia
* No allergy or hypersensitivity to heparin, tinzaparin sodium, pork products, sulfite, or benzyl alcohol
* No uncontrolled severe intercurrent illness, including ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* No uncontrolled arterial hypertension, history of gastrointestinal ulceration, and/or bleeding in the past 4 weeks
* No diabetic retinopathy or history of retinal hemorrhage
* Not pregnant or nursing
* HIV-positive patients are allowed

PRIOR CONCURRENT THERAPY:

* No treatment with anticoagulation lasting > 1 month in the past 6 months
* No anticoagulation, including treatment with a low molecular weight heparin, at any time within the past month
* More than 4 weeks since prior surgery, radiation therapy, immunotherapy, or chemotherapy
* Recovered from prior therapy
* No other concurrent investigational agents
* No other concurrent anticoagulation therapy, including oral anticoagulants, thrombolytic agents, or any form of heparin

  * Concurrent antiplatelet agents allowed
* No spinal or epidural puncture, anesthesia, or post-operative indwelling epidural catheters within the past 48 hours
* No other concurrent anticancer agents or therapies
* No concurrent sex hormones except for postmenopausal hormone replacement
* No concurrent chemotherapy or immunotherapy
* No concurrent palliative radiotherapy
* Concurrent urgent use of corticosteroids allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2005-12; Primary Completion 2007-02 (Estimated)

PRIMARY OUTCOMES:
Blood markers or coagulation as measured by plasma prothrombin F1.2, thrombin-antithrombin complexes, and D-dimers at 2 weeks, 2 months and 6 months

SECONDARY OUTCOMES:
Blood markers of angiogenesis as measured by serum vascular endothelial growth factor (VEGF) and basic fibroblast growth factor (bFGF) at 2 weeks, 2 months, and 6 months
Venous thromboembolism as measured by clinical evaluation at 6 months
Progression free survival as measured by clinical evaluation at 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L. Ornstein, MD, Study Chair — Yale University
Locations (3):
- United States (3):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont